CLINICAL TRIAL: NCT01538433
Title: A Survey of Factors Affecting an Early or Delayed Diagnosis of IgA Nephropathy: an Observational Study
Brief Title: A Survey of Factors Affecting an Early or Delayed Diagnosis of IgA Nephropathy
Status: Completed | Type: Observational
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Wei Shi, Prof., Guangdong Provincial People's Hospital
Other Study IDs: GGH201107
Record Dates: First submitted 2012-02-19; First posted 2012-02-24 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2013-08

CONDITIONS: IgA Nephropathy
Keywords: diagnosis; IgA nephropathy
MeSH Terms: conditions — Glomerulonephritis, IGA; Disease

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- biopsy-proven IgA nephropathy

SUMMARY:
This is a survey of factors which affect a pathologically defined early or delayed diagnosis of IgA nephropathy in Guangdong General Hospital, Guangzhou, China. An early or delayed diagnosis of IgA nephropathy is pathologically defined using the recently published Oxford classification of IgA nephropathy. The factors to be surveyed include health examination including urine test, socioeconomic status of patients including education,etc.

ELIGIBILITY:
Inclusion Criteria:

* biopsy-proven IgA Nephropathy patients in Guangdong General Hospital, Guangzhou,China

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The consecutive biopsy-proven IgAN patients in Guangdong General Hospital, Guangzhou,China
Sampling Method: Probability Sample
Enrollment: 603 (Actual)
Dates: Start 2012-02; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Factors potentially affecting an early or delayed diagnosis of IgA Nephropathy | Before the biopsy

SECONDARY OUTCOMES:
Glomerular filtration rate(GFR) decline rate or reaching end-stage renal disease (ESRD) or doubling of serum creatinine | after the biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Wei Shi, MD, PhD, Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Nephrology Department,Guangdong General Hospital, Guangzhou, Guangdong, China